CLINICAL TRIAL: NCT03834077
Title: The Effect of Tissue Flossing in Patients With Tennis Elbow
Brief Title: Tissue Flossing in Tennis Elbow Patients
Acronym: FLOSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Vice Dean, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ujaenflossing
Record Dates: First submitted 2019-02-04; First posted 2019-02-07 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Tennis Elbow
Keywords: physiotherapy
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be allocated to intervention (flossing) or control group (conventional physiotherapy) using a randomized list of allocated numbers generated by a computer program. Opaque envelope will contain the patients allocation while outcome assessors, care provider and principal investigator will be blinded to the allocation process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tissue flossing (Experimental): Conventional physiotherapy consisted in electrotherapy and stretching in addition to tissue flossing.
  Interventions: Other: Tissue flossing
- Placebo comparator (Placebo Comparator): Conventional physiotherapy consisted in electrotherapy and stretching in addition with tissue flossing without tension.
  Interventions: Other: Placebo comparator

INTERVENTIONS:
Other: Tissue flossing — Electrotherapy (transcutaneous electrical nerve stimulation) and Ultrasound in addition to tissue flossing.
  Arms: Tissue flossing
Other: Placebo comparator — Conventional physiotherapy in addition to flossing without tension
  Arms: Placebo comparator

SUMMARY:
The aim of the present intervention is to determine the effectiveness of the application of tissue flossing in patients with tennis elbow

DETAILED DESCRIPTION:
The application of tissue flossing has been deemed to provide beneficial results in patients with ankle range of motion limitation. Although, tissue flossing is widely extended among athletes due to its effectiveness in pain, function and range of motion, the evidence is limited.

The aim of the present protocol is to determine the effectiveness of tissue flossing in patients with tennis elbow.

ELIGIBILITY:
Inclusion Criteria:

* Elbow pain for at least 6 weeks and satisfy the widely accepted diagnostic criteria of lateral epicondylalgia.
* Diagnostic criteria are pain over the lateral humeral epicondyle that is provoked by gripping activities.
* Reduced grip strength and increased sensitivity to manual palpation over the lateral epicondyle.
* Pain with stretching or contraction of the wrist extensor muscles.

Exclusion Criteria:

* Upper limb fractures, surgery or concomitant disease.
* Red flags presence.
* Mental disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-03-28 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Patient-related Tennis Elbow Questionnaire change | At baseline, after 1 week and after 4 week.
  Self reported questionnaire ranged from 0 to 150 with greater scores associated with severe disability.

SECONDARY OUTCOMES:
Numeric rating scale change | At baseline, after 1 week and after 4 week.
  10 point rating scale of pain where 0 is associated with no pain and 10 with greatest pain.
Pressure Pain Threshold change | At baseline, after 1 week and after 4 week.
  Determine the pain free pression with a validated instrument

CONTACTS AND LOCATIONS:
Overall Officials: David Cruz-Diaz, PhD, Principal Investigator — University of Jaen
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: Undecided
This intervention could be beneficial to support or refuse the use of tissue flossing.